CLINICAL TRIAL: NCT03546413
Title: Follow up of Learning Early About Peanut Allergy (LEAP) Participants and Their Families: LEAP Trio (ITN070AD)
Brief Title: Follow up of LEAP Participants and Their Families
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: DAIT ITN070AD; LEAP Trio (Other: Immune Tolerance Network); NIAID CRMS ID#: 38498 (Other: DAIT NIAID)
Record Dates: First submitted 2018-04-17; First posted 2018-06-06 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Peanut Allergy
Keywords: food; peanut; allergy; prevention
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be collected for peripheral blood mononuclear cell (PBMC) isolation and sent to the Immune Tolerance Network (ITN) designated core laboratory for processing using ITN approved standard operating procedures (SOPs) for PBMC separation and aliquoting. These cells will be available for future studies such as immunosequencing and functional studies when remaining cell numbers are sufficient to make these assays technically feasible. DNA will be collected for genetic analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- LEAP Participants: Peanut Avoidance: Participants of the LEAP study who enrolled in the LEAP Trio study and were originally randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study.
- LEAP Participants: Peanut Consumption: Participants of the LEAP study who enrolled in the LEAP Trio study and were originally randomized to the Peanut Consumption treatment arm upon entry into the LEAP study.
- Younger Siblings: Peanut Avoidance: Participants enrolled in the LEAP Trio study who are younger siblings of a LEAP Participant who was randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study.
- Younger Siblings: Peanut Consumption: Participants enrolled in the LEAP Trio study who are younger siblings of a LEAP Participant who was randomized to the Peanut Consumption treatment arm upon entry into the LEAP study.
- Older Siblings: Peanut Avoidance: Participants enrolled in the LEAP Trio study who are older siblings of a LEAP Participant who was randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study.
- Older Siblings: Peanut Consumption: Participants enrolled in the LEAP Trio study who are older siblings of a LEAP Participant who was randomized to the Peanut Consumption treatment arm upon entry into the LEAP study.
- Parents: Peanut Avoidance: Participants enrolled in the LEAP Trio study who are parents of a LEAP Participant who was randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study.
- Parents: Peanut Consumption: Participants enrolled in the LEAP Trio study who are parents of a LEAP Participant who was randomized to the Peanut Consumption treatment arm upon entry into the LEAP study.

SUMMARY:
This prospective, cross-sectional study was designed to improve understanding of how early-life introduction of peanuts may promote the maintenance of tolerance in adolescence and will serve as an additional safety evaluation of the original nutritional intervention.

DETAILED DESCRIPTION:
Background: Food allergies and specifically peanut allergy (PA) are increasingly common conditions and are an important public health concern. Dietary avoidance of peanut in early life has been recommended in many countries. However, there is evidence that the prevalence of PA is decreased in countries where children are fed peanut beginning at an early age.

The LEAP (Learning Early About Peanut allergy) Study (Protocol ITN032AD, NCT00329784) demonstrated that the early consumption of peanut in high-risk infants successfully reduced the prevalence of peanut allergy at five years of age when compared to peanut avoidance. The LEAP-On Study (Protocol ITN049AD, NCT01366846) was a follow-on study to LEAP and demonstrated that children who consumed peanut in the LEAP study remained protected against developing peanut allergy after cessation of peanut consumption for a period of 12 months.

This LEAP Trio cohort study, a longer-term follow-up of the LEAP study participants, assessed whether the benefits of regular early-life peanut consumption are maintained over many years when peanut consumption is ad libitum (in the amount and frequency chosen by the individual participant).

The three cohorts in LEAP-Trio include:

* LEAP Participants (NCT00329784, NCT01366846)
* their Siblings and
* their Parents

The study began on July 5, 2018, with data collection continuing until August 31, 2022. This allowed for the enrollment of former LEAP participants aged 12 years.:

• The enrollment phase was 217 weeks (4 years, 2 months).

--The LEAP siblings and parents were enrolled concurrently with the LEAP participant.

• Study participation was defined as a single visit (Visit 144 months); however, more than one clinic appointment might have been required to complete all assessments and were required to be completed within 8 weeks of the in-person visit. Due to COVID-19, telephone visits were undertaken when participants were not able to or did not wish to come into the clinic or have a home visit. The visit window did not apply to the telephone visit. Participants who underwent a telephone visit were invited to subsequently undergo an in-person clinic visit or home visit.

Participant assessments included general medical, -dietary, -allergy (including but not limited to oral peanut food challenges for former LEAP participants and their siblings), and mechanistic assessments (involving the collection of biological specimens, a blood draw, skin prick testing, as examples, to explore hypotheses related to potential mechanisms of peanut allergy).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - LEAP Participants:

* Participation in LEAP;
* At least 9.5 years of age
* Willingness to participate in at least one study data collection (i.e. questionnaire, skin pricking testing, or blood draw) procedure; and
* Assent by child and informed consent by parent or legal guardian.

Inclusion Criteria - LEAP Siblings:

* Sibling of LEAP participant;
* Willingness to participate in at least one study data collection (i.e. questionnaire, skin pricking testing, or blood draw); and
* Assent by child and informed consent by parent or legal guardian if child is younger than 16; siblings aged 16 and over will provide their own consent.

Inclusion Criteria - LEAP Parents:

* Biological parent of LEAP participant;
* Willingness to participate in at least one study data collection (i.e. questionnaire, skin pricking testing, or blood draw); and
* Informed consent (for participants only returning a Questionnaire, informed consent will be implied).

Exclusion Criteria:

* There are no exclusion criteria for LEAP Participants, LEAP Siblings, LEAP Parents

Min Age: 0 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Original Learning Early About Peanut (LEAP) allergy study participants (NCT00329784): at high risk for peanut allergy, given the presence of severe eczema, egg allergy, or both
  * Siblings of LEAP participants
  * Parents of LEAP participants
Sampling Method: Non-Probability Sample
Enrollment: 1868 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Lack, MD, Study Chair — Evelina Children's Hospital, Guy's and St. Thomas's NHS Foundation Trust
Locations (1):
- Evelina London Children's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Background] Sever ML, Calatroni A, Roberts G, du Toit G, Bahnson HT, Radulovic S, Larson D, Byron M, Santos AF, Huffaker MF, Wheatley LM, Lack G. Developing a Prediction Model for Determination of Peanut Allergy Status in the Learning Early About Peanut Allergy (LEAP) Studies. J Allergy Clin Immunol Pract. 2023 Jul;11(7):2217-2227.e9. doi: 10.1016/j.jaip.2023.04.032. Epub 2023 May 3. PMID 37146884
- [Derived] Du Toit G, Huffaker MF, Radulovic S, Feeney M, Fisher HR, Byron M, Dunaway L, Calatroni A, Johnson M, Foong RX, Marques-Mejias A, Bartha I, Basting M, Brough HA, Baloh C, Laidlaw TM, Bahnson HT, Roberts G, Plaut M, Wheatley LM, Lack G; Immune Tolerance Network LEAP-Trio Trial Team. Follow-up to Adolescence after Early Peanut Introduction for Allergy Prevention. NEJM Evid. 2024 Jun;3(6):EVIDoa2300311. doi: 10.1056/EVIDoa2300311. Epub 2024 May 28. PMID 38804779
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — https://www.immunetolerance.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This longer-term follow-up of the LEAP study participants assessed whether the benefits of regular early-life peanut consumption are maintained over many years when followed by consumption of peanut ad lib, in the amount and at frequency chosen by the individual participant.
  The LEAP siblings and parents cohorts were also enrolled concurrently with the LEAP participant cohort.
Period: Overall Study
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Started | 253 | 255 | 193 | 191 | 76 | 91 | 400 | 409
Completed | 253 | 255 | 193 | 191 | 76 | 91 | 400 | 409
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All LEAP Trio enrolled participants
Groups:
- LEAP Participants: Peanut Avoidance: Participants of the LEAP study who enrolled in the LEAP Trio study and were originally randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study. Target accrual is 316.
- LEAP Participants: Peanut Consumption: Participants of the LEAP study who enrolled in the LEAP Trio study and were originally randomized to the Peanut Consumption treatment arm upon entry into the LEAP study. Target accrual is 314
- Younger Siblings: Peanut Avoidance: Participants enrolled in the LEAP Trio study who are younger siblings of a LEAP Participant who was randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study. Target accrual is 222.
- Younger Siblings: Peanut Consumption: Participants enrolled in the LEAP Trio study who are younger siblings of a LEAP Participant who was randomized to the Peanut Consumption treatment arm upon entry into the LEAP study. Target accrual is 207.
- Older Siblings: Peanut Avoidance: Participants enrolled in the LEAP Trio study who are older siblings of a LEAP Participant who was randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study. Target accrual is 153.
- Older Siblings: Peanut Consumption: Participants enrolled in the LEAP Trio study who are older siblings of a LEAP Participant who was randomized to the Peanut Consumption treatment arm upon entry into the LEAP study. Target accrual is 164.
- Parents: Peanut Avoidance: Participants enrolled in the LEAP Trio study who are parents of a LEAP Participant who was randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study Target accrual is 474.
- Parents: Peanut Consumption: Participants enrolled in the LEAP Trio study who are parents of a LEAP Participant who was randomized to the Peanut Consumption treatment arm upon entry into the LEAP study. Target accrual is 471.
- Total: Total of all reporting groups
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption | Total
Number analyzed (Participants) | 253 | 255 | 193 | 191 | 76 | 91 | 400 | 409 | 1868
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.0 (1.15) | 12.9 (1.17) | 9.6 (2.29) | 9.8 (2.26) | 17.1 (3.48) | 17.3 (3.51) | 47.1 (4.97) | 47.7 (5.22) | 27.6 (17.82)
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 253 | 255 | 193 | 191 | 57 | 65 | 0 | 0 | 1014
  Between 18 and 65 Years | 0 | 0 | 0 | 0 | 19 | 26 | 398 | 407 | 850
  >65 Years | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 90 | 120 | 93 | 83 | 36 | 50 | 241 | 249 | 962
  Gender: Male | 162 | 135 | 100 | 108 | 40 | 41 | 158 | 160 | 904
  Gender: Undifferentiated or Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 200 | 181 | 161 | 140 | 62 | 72 | 340 | 325 | 1481
  Race: Black | 13 | 16 | 7 | 9 | 8 | 4 | 24 | 27 | 108
  Race: Asian | 8 | 9 | 3 | 6 | 3 | 4 | 19 | 22 | 74
  Race: Chinese, Middle Eastern, or Other Ethnic Group | 3 | 9 | 3 | 8 | 0 | 1 | 8 | 14 | 46
  Race: More than one race | 27 | 38 | 19 | 23 | 3 | 9 | 7 | 12 | 138
  Race: Unknown or Not Reports | 2 | 2 | 0 | 5 | 0 | 1 | 2 | 9 | 21
Region of Enrollment [Number; unit: participants]
  United Kingdom | 253 | 255 | 193 | 191 | 76 | 91 | 400 | 409 | 1868

OUTCOME MEASURES:

1. Primary Outcome: Percentage of LEAP Participants With Peanut Allergy
Description: Peanut allergy status at LEAP Trio Visit 144 was determined by peanut challenge where possible. Participants who met criteria for peanut oral allergy syndrome in the absence of primary peanut allergy were not considered peanut allergic. Individuals who reported consuming at least 2 g of peanut protein without reaction on at least one occasion in the last year were considered peanut tolerant. If oral challenge was not possible and participants did not meet the above criteria for tolerance, peanut allergy status was determined by an internally and externally validated novel peanut allergy prediction model using data for peanut wheal size (mm), peanut specific IgE (kU/L), Ara h1 (kU/L), Ara h2 (kU/L) and Ara h3 (kU/L)
Time Frame: Assessments were performed on consented LEAP Participants at the time of the LEAP Participant's Visit 144 (when the LEAP Study (NCT00329784) Participant was approximately 12 years old (age approximately 144 months)).
Population: All LEAP Trio participants in the LEAP Participant cohort for whom data was available to make a determination of peanut allergy status at LEAP Trio Visit 144.
Measure: Number; unit: Percentage of Participants
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 246 | 251 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of Participants
  Allergic | 15.4 | 4.4 |  |  |  |  |  |
  Tolerant | 84.6 | 95.6 |  |  |  |  |  |
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test for equivalence between the groups; Test type: Superiority; p < 0.001, Regression, Logistic — This is the calculated p-value

2. Primary Outcome: Percentage of Younger Siblings With Peanut Sensitization
Description: Peanut sensitization in the siblings of the LEAP Participants was defined as meeting at least one of the following criteria:
  Specific-IgE ≥0.35 kU/L or Specific-IgE to individual peanut component Ara h2 ≥0.1 kU/L, or Skin prick test wheal to peanut ≥3mm
Time Frame: Assessments were performed on consented siblings at the time of the LEAP Participant's Visit 144 (when the LEAP Study (NCT00329784) Participant was approximately 12 years old (age approximately 144 months)).
Population: Siblings of the LEAP Participants who met the following criteria: Younger Siblings who were enrolled in LEAP Trio, resided in the home of the LEAP Participant during the LEAP Study (NCT00329784), and had results at LEAP Trio Visit 144 for peanut specific IgE, specific-IgE to individual peanut component Ara h2, or skin prick test wheal to peanut.
Measure: Number; unit: Percentage of Particpants
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 0 | 0 | 130 | 135 | 0 | 0 | 0 | 0
Percentage of Particpants
  Sensitized |  |  | 20.0 | 30.4 |  |  |  |
  Not Sensitized |  |  | 80.0 | 69.6 |  |  |  |
Statistical Analysis 1: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test for equivalence between the groups; Test type: Superiority — A logistic regression model was used with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for siblings who are in the same family unit; p = 0.055, Regression, Logistic

3. Secondary Outcome: Average Weekly Peanut Protein Consumption of LEAP Participants, Younger Siblings, Older Siblings and Parents
Description: At LEAP Trio Visit 144, participants were asked to provide responses to questions about their peanut protein consumption. Responses obtained at LEAP Trio Visit 144 were based on the recollection of peanut consumption during the 4 weeks prior to the LEAP Trio study Visit 144.
Time Frame: Assessments were performed on consented LEAP Participants and family members at the time of the LEAP Participant's Visit 144 (when the LEAP Study (NCT00329784) Participant was approximately 12 years old (age approximately 144 months)).
Population: All participants in LEAP Trio who provided a response to the question of average weekly peanut protein consumption in the 4 weeks prior to LEAP Trio Visit 144.
Measure: Median (Full Range); unit: Grams
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 251 | 253 | 188 | 187 | 76 | 91 | 398 | 400
Grams | 0.0 [0.0 to 92.1] | 5.2 [0.0 to 120.0] | 0.7 [0.0 to 63.4] | 2.6 [0.0 to 97.0] | 1.4 [0.0 to 49.3] | 1.3 [0.0 to 120.7] | 3.6 [0.0 to 82.2] | 5.3 [0.0 to 130.0]
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — This is the calculated p-value
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — A linear regression model was used on the log of the peanut consumption with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for siblings who are in the same family unit; p < 0.001, Regression, Linear — This is the calculated p-value
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 3, analysis 2]; p = 0.939, Regression, Linear
Statistical Analysis 4: Comparison: Parents: Peanut Avoidance vs Parents: Peanut Consumption; Test type: Superiority — A linear regression model was used on the log of the peanut consumption with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for parents who are in the same family unit; p = 0.002, Regression, Linear

4. Secondary Outcome: Peanut Skin Prick Test Wheal Size for LEAP Participants, Younger Siblings, Older Siblings and Parents
Description: Skin prick tests were performed to assess participants for potential peanut allergy, select food allergens, and select aeroallergens
Time Frame: as for outcome 3
Population: All participants in LEAP Trio for whom data was available for peanut skin prick test wheal at LEAP Trio Visit 144.
Measure: Median (Full Range); unit: Millimeters
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 213 | 225 | 161 | 165 | 64 | 73 | 331 | 342
Millimeters | 0.0 [0.0 to 30.0] | 0.0 [0.0 to 22.0] | 0.0 [0.0 to 15.0] | 0.0 [0.0 to 16.0] | 0.0 [0.0 to 5.0] | 0.0 [0.0 to 13.0] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 7.0]
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p = 0.131, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — A linear regression model was used on the log of peanut skin prick test with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for siblings who are in the same family unit; p = 0.208, Regression, Linear
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Superiority — A linear regression model was used on the log of peanut skin prick with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for siblings who are in the same family unit; p = 0.587, Regression, Linear
Statistical Analysis 4: Comparison: Parents: Peanut Avoidance vs Parents: Peanut Consumption; Test type: Superiority — A linear regression model was used on the log of peanut skin prick with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for parents who are in the same family unit; p = 0.268, Regression, Linear

5. Secondary Outcome: Peanut Specific-IgE Measurements for the LEAP Participants, Younger Siblings, Older Siblings, and Parents
Description: Participants had blood draws to assess specific-IgE measurements to peanut, select food allergens and select aeroallergens
Time Frame: as for outcome 3
Population: All participants in LEAP Trio for whom data was available for peanut specific IgE at LEAP Trio Visit 144
Measure: Median (Full Range); unit: kU/Liter
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 210 | 221 | 157 | 147 | 61 | 72 | 349 | 360
kU/Liter | 0.2 [0.1 to 481.0] | 0.2 [0.1 to 188.0] | 0.1 [0.1 to 891.0] | 0.1 [0.1 to 707.0] | 0.1 [0.1 to 6.5] | 0.1 [0.1 to 44.4] | 0.1 [0.1 to 8.5] | 0.1 [0.1 to 12.5]
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p = 0.985, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — A linear regression model was used on the log of peanut specific IgE with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for siblings who are in the same family unit; p = 0.371, Regression, Linear
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 5, analysis 2]; p = 0.483, Regression, Linear
Statistical Analysis 4: Comparison: Parents: Peanut Avoidance vs Parents: Peanut Consumption; Test type: Superiority — A linear regression model was used on the log of peanut specific IgE with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for parents who are in the same family unit; p = 0.643, Regression, Linear

6. Secondary Outcome: SCORAD Score for the Eczema Severity in LEAP Participants, Younger Siblings and Older Siblings
Description: Eczema severity was assessed using a modified Scoring Atopic Dermatitis (SCORAD) assessment. The range of the SCORAD is 0-103. A score of 0 indicates no eczema, scores between 0 and 15 indicate mild eczema, scores between 15 and 40 indicate moderate eczema, and scores greater than 40 indicate severe eczema.
Time Frame: as for outcome 3
Population: All participants in LEAP Trio in the LEAP Participants, Younger Siblings and Older Siblings cohorts for whom data was available for the SCORAD evaluation at LEAP Trio Visit 144
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 215 | 223 | 160 | 167 | 64 | 70 | 0 | 0
Units on a scale | 0.0 [0.0 to 65.8] | 0.0 [0.0 to 161.0] | 0.0 [0.0 to 63.1] | 0.0 [0.0 to 77.1] | 0.0 [0.0 to 37.0] | 0.0 [0.0 to 56.2] |  |
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p = 0.225, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — A linear regression model was used on the log of SCORAD with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for siblings who are in the same family unit; p = 0.857, Regression, Linear
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 6, analysis 2]; p = 0.870, Regression, Linear

7. Secondary Outcome: Percentage of LEAP Participants, Younger Siblings, Older Siblings, and Parents With Eczema
Description: Participants were classified as having eczema using standard methodology. Participants were assessed for eczema using a modified Scoring Atopic Dermatitis System (SCORAD) and using participant report of a history of eczema. The range of the SCORAD is 0-103. A score of 0 indicates no eczema, scores between 0 and 15 indicate mild eczema, scores between 15 and 40 indicate moderate eczema, and scores greater than 40 indicate severe eczema.
Time Frame: as for outcome 3
Population: All participants in LEAP Trio in the Intent-to-Treat population: participants with at least one assessment completed at LEAP Trio Visit 144.
Measure: Number; unit: Percentage of Participants
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 253 | 255 | 193 | 191 | 76 | 91 | 400 | 409
Percentage of Participants
  Has Eczema | 49.4 | 51.4 | 24.4 | 31.9 | 25.0 | 29.7 | 17.3 | 19.6
  Does Not Have Eczema | 50.6 | 48.6 | 75.6 | 68.1 | 75.0 | 70.3 | 82.7 | 80.4
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p = 0.658, Regression, Logistic
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.100, Regression, Logistic
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.502, Regression, Linear
Statistical Analysis 4: Comparison: Parents: Peanut Avoidance vs Parents: Peanut Consumption; Test type: Superiority — A logistic regression model was used with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for parents who are in the same family unit; p = 0.397, Regression, Linear

8. Secondary Outcome: Percentage of LEAP Participants, Younger Siblings, Older Siblings, and Parents With Asthma
Description: Participants were classified as having asthma if they meet at least one of the following definitions:
  1. Participant report of cough, wheeze, or shortness of breath that was responsive to therapy with bronchodilators on two or more occasions in the previous 24 months; or required one visit to a physician in the previous 24 months; or occurred during the night, during early morning, or upon exercising in the intervals between exacerbations at any time in the previous 12 months.
  2. Participant report of an asthma diagnosis with current use of asthma medications (short-acting beta-agonist or controller)
  3. Participant report of transient wheeze on exposure to a suspected allergen with confirmatory allergy tests
Time Frame: as for outcome 3
Population: All participants in LEAP Trio for whom data was available to make a determination of asthma status at LEAP Trio Visit 144.
Measure: Number; unit: Percentage of Participants
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 248 | 253 | 186 | 189 | 76 | 88 | 400 | 409
Percentage of Participants
  Has Asthma | 33.5 | 31.6 | 15.1 | 11.1 | 11.8 | 22.7 | 8.5 | 11.2
  Does Not Have Asthma | 66.5 | 68.4 | 84.9 | 88.9 | 88.2 | 77.3 | 91.5 | 88.8
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p = 0.659, Regression, Logistic
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.260, Regression, Logistic
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.075, Regression, Linear
Statistical Analysis 4: Comparison: Parents: Peanut Avoidance vs Parents: Peanut Consumption; Test type: Superiority — [test comment as in outcome 7, analysis 4]; p = 0.192, Regression, Logistic

9. Secondary Outcome: Percentage of LEAP Participants, Younger Siblings, Older Siblings, and Parents With Perennial Rhinitis
Description: Participants were considered to have perennial rhinitis if they demonstrated a sensitization to the aeroallergen and clinical history of rhinoconjunctivitis symptoms experienced when exposed to the relevant allergen. Sensitization to the relevant allergen was defined as:
  1. Allergen specific IgE ≥ 0.35 kU/L, or
  2. Skin prick test wheal size to allergen ≥ 3 mm.
Time Frame: as for outcome 3
Population: All participants in LEAP Trio for whom data was available to make a determination of perennial rhinitis status at LEAP Trio Visit 144.
Measure: Number; unit: Percentage of Participants
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 253 | 255 | 193 | 191 | 76 | 91 | 400 | 409
Percentage of Participants
  Has Perennial Rhinitis | 44.3 | 42.7 | 16.1 | 17.3 | 17.1 | 26.4 | 18.0 | 20.0
  Does Not Have Perennial Rhinits | 55.7 | 57.3 | 83.9 | 82.7 | 82.9 | 73.6 | 82.0 | 80.0
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p = 0.729, Regression, Logistic
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.750, Regression, Logistic
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.155, Regression, Logistic
Statistical Analysis 4: Comparison: Parents: Peanut Avoidance vs Parents: Peanut Consumption; Test type: Superiority — [test comment as in outcome 7, analysis 4]; p = 0.458, Regression, Logistic

10. Secondary Outcome: Percentage of LEAP Participants, Younger Siblings, Older Siblings and Parents With Seasonal Rhinitis
Description: Participants were considered to have seasonal rhinitis if they demonstrated a sensitization to a seasonal aeroallergen and clinical history of rhinoconjunctivitis symptoms experienced when exposed to the allergen during the relevant season. Sensitization to the relevant allergen was defined as:
  1. Allergen specific IgE ≥ 0.35 kU/L, or
  2. Skin prick test wheal size to allergen ≥ 3 mm
Time Frame: as for outcome 3
Population: All participants in LEAP Trio for whom data was available to make a determination of seasonal rhinitis status at LEAP Trio Visit 144.
Measure: Number; unit: Percentage of Participants
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 253 | 255 | 193 | 191 | 76 | 91 | 400 | 409
Percentage of Participants
  Has Seasonal Rhinitis | 49.0 | 53.3 | 18.7 | 22.5 | 25.0 | 29.7 | 24.5 | 23.5
  Does Not Have Seasonal Rhinitis | 51.0 | 46.7 | 81.3 | 77.5 | 75.0 | 70.3 | 75.5 | 76.5
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p = 0.330, Regression, Logistic
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.351, Regression, Logistic
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.502, Regression, Logistic
Statistical Analysis 4: Comparison: Parents: Peanut Avoidance vs Parents: Peanut Consumption; Test type: Superiority; p = 0.732, Regression, Logistic — A logistic regression model was used with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for parents who are in the same family unit

11. Secondary Outcome: Percentage of LEAP Younger Siblings, Older Siblings and Parents With Peanut Allergy
Description: as for outcome 1
Time Frame: Assessments were performed on consented family members at the time of the LEAP Participant's Visit 144 (when the LEAP Study (NCT00329784) Participant was approximately 12 years old (age approximately 144 months)).
Population: All participants in LEAP Trio in the Younger Siblings, Older Siblings and Parents cohorts for whom data was available to make a determination of peanut allergy status at LEAP Trio Visit 144. Results for peanut allergy of LEAP Participants are displayed in Primary Outcome Measure #1
Measure: Number; unit: Percentage of Participants
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 0 | 0 | 189 | 187 | 74 | 89 | 397 | 407
Percentage of Participants
  Allergic |  |  | 4.8 | 8.0 | 0.0 | 2.2 | 0.3 | 0.0
  Tolerant |  |  | 95.2 | 92.0 | 100.0 | 97.8 | 99.7 | 100.0
Statistical Analysis 1: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.202, Regression, Logistic
Statistical Analysis 2: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Other; Regression, Logistic; A logistic regression model was used with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for siblings who are in the same family unit. However, the logistic regression model was unable to converge due to the low percentage of allergic participants in older siblings
Statistical Analysis 3: Comparison: Parents: Peanut Avoidance vs Parents: Peanut Consumption; Test type: Other; Regression, Logistic; A logistic regression model was used with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for parents who are in the same family unit. However, the logistic regression model was unable to converge due to the low percentage of allergic participants in parents

12. Secondary Outcome: Percentage of LEAP Participants, Younger Siblings and Older Siblings With at Least One Peanut-related Adverse Event
Description: Peanut-related adverse events were reported from reactions experienced during or within 30 days after the LEAP Trio Visit 144 peanut oral food challenge (peanut OFC)
Time Frame: Within 30 days after peanut OFC performed on consented LEAP Participants and family members at the time of the LEAP Participant's Visit 144 (when the LEAP Study (NCT00329784) Participant was approximately 12 years old (age approximately 144 months)).
Population: All participants in LEAP Trio in the LEAP Participants, Younger Siblings and Older Siblings cohorts in the Intent-to-Treat population: participants with at least one assessment completed at LEAP Trio Visit 144. The peanut oral food challenge was not performed in Parents.
Measure: Number; unit: Percentage of Participants
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | Parents: Peanut Avoidance | Parents: Peanut Consumption
Number analyzed (Participants) | 253 | 255 | 193 | 191 | 76 | 91 | 0 | 0
Percentage of Participants
  Had Peanut-related AE | 5.9 | 2.0 | 2.6 | 1.6 | 0.0 | 0.0 |  |
  Did Not Have Peanut-related AE | 94.1 | 98.0 | 97.4 | 98.4 | 100.0 | 100.0 |  |
Statistical Analysis 1: Comparison: LEAP Participants: Peanut Avoidance vs LEAP Participants: Peanut Consumption; Test type: Superiority; p = 0.029, Regression, Logistic
Statistical Analysis 2: Comparison: Younger Siblings: Peanut Avoidance vs Younger Siblings: Peanut Consumption; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.489, Regression, Logistic
Statistical Analysis 3: Comparison: Older Siblings: Peanut Avoidance vs Older Siblings: Peanut Consumption; Test type: Other; Regression, Logistic; A logistic regression model was used with a fixed effect comparing the Avoidance and Consumption cohorts and a random effect to account for siblings who are in the same family unit. However, the model was unable to converge due to the low percentage of peanut-related adverse events in older siblings

ADVERSE EVENTS:
Time Frame: Consents and assessments were performed on LEAP Participants and family members at the time of the LEAP Participant's Visit 144 (when the LEAP Study (NCT00329784) Participant was approximately 12 years old (age approximately 144 months)). AEs were collected during each study visit and up to 30 days after each visit, or until the event was resolved, whichever came first (up to a maximum of 2 visits, and maximum of 38 months in the study). Original 8-week window was extended due to COVID-19.
Description: This is a trial with a single planned study visit at LEAP Trio Visit 144. As a cross-sectional study, it did not aim to capture disease or therapy-related adverse events over time. The principal aim was to capture adverse events that may be related to study procedures.
Groups:
- LEAP Parents: Peanut Avoidance; LEAP Parents: Peanut Consumption: Participants enrolled in the LEAP Trio study who are parents of a LEAP Participant who was randomized to the Peanut Avoidance treatment arm upon entry into the LEAP study
Arm/Group | LEAP Participants: Peanut Avoidance | LEAP Participants: Peanut Consumption | Younger Siblings: Peanut Avoidance | Younger Siblings: Peanut Consumption | Older Siblings: Peanut Avoidance | Older Siblings: Peanut Consumption | LEAP Parents: Peanut Avoidance | LEAP Parents: Peanut Consumption
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/255 | 0/193 | 0/191 | 0/76 | 0/91 | 0/400 | 0/409
Serious Adverse Events (participants affected / at risk) | 1/253 | 0/255 | 2/193 | 0/191 | 0/76 | 0/91 | 0/400 | 0/409
Other Adverse Events (participants affected / at risk) | 20/253 | 6/255 | 3/193 | 5/191 | 0/76 | 0/91 | 0/400 | 0/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEAP Participants: Peanut Avoidance (N=253) | LEAP Participants: Peanut Consumption (N=255) | Younger Siblings: Peanut Avoidance (N=193) | Younger Siblings: Peanut Consumption (N=191) | Older Siblings: Peanut Avoidance (N=76) | Older Siblings: Peanut Consumption (N=91) | LEAP Parents: Peanut Avoidance (N=400) | LEAP Parents: Peanut Consumption (N=409)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEAP Participants: Peanut Avoidance (N=253) | LEAP Participants: Peanut Consumption (N=255) | Younger Siblings: Peanut Avoidance (N=193) | Younger Siblings: Peanut Consumption (N=191) | Older Siblings: Peanut Avoidance (N=76) | Older Siblings: Peanut Consumption (N=91) | LEAP Parents: Peanut Avoidance (N=400) | LEAP Parents: Peanut Consumption (N=409)
Injection site pruritus (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 13 (13) | 5 (5) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03546413/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT03546413/SAP_001.pdf